CLINICAL TRIAL: NCT01108094
Title: Pilot Biomarker Trial to Evaluate the Efficacy of Itraconazole in Patients With Basal Cell Carcinomas
Brief Title: Pilot Biomarker Trial to Evaluate the Efficacy of Itraconazole in Patients w/ Basal Cell Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17365; SU-04162010-5722 (Other: Stanford University); SKIN0004-TX (Other: OnCore)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Basal Cell Carcinoma (BCC); Skin Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A - Itraconazole 400 mg (Experimental): Oral itraconazole 400 mg as 200 mg twice daily, for 1 month, stratified by prior vismodegib history
  Interventions: Drug: Itraconazole
- Cohort B - Itraconazole 200 mg (Experimental): Oral itraconazole 200 mg as 100 mg twice daily, for up to 3 months
  Interventions: Drug: Itraconazole
- Untreated Control (No Intervention): Patients otherwise eligible but unwilling to take itraconazole were enrolled onto the control arm of the study and received no treatment

INTERVENTIONS:
Drug: Itraconazole — * Cohort A: oral itraconazole 400 mg as 200 mg twice daily; for 1 month
  * Cohort B: oral itraconazole 200 mg as 100 mg twice daily; for up to 3 months
  Other Names: Sporanox
  Arms: Cohort A - Itraconazole 400 mg; Cohort B - Itraconazole 200 mg

SUMMARY:
Basal cell carcinomas (BCCs) are the most common human cancer in the US and affect over 1 million people. There is no effective drug to prevent basal cell carcinomas of the skin.

We hope to learn if an oral anti-fungal drug, itraconazole, might inhibit a marker of proliferation and a biomarker (tumor signaling pathway) of BCC development.

Itraconazole is an FDA-approved drug for the treatment of fungal infections of the skin, and has been used for the past 25 years with relatively few side effects. It has been shown in mice to reduce a BCC biomarker and to reduce growth of BCCs.

Thus, it may reduce BCC growth in humans.

DETAILED DESCRIPTION:
Participants with at least one BCC tumor measuring 4 mm or greater in diameter will be enrolled onto 1 of 2 treatment cohorts to receive oral itraconazole.

* Cohort A - 400 mg itraconazole (as 200 mg twice daily for 30 days), stratified by:

  * Cohort A1 - Participants are vismodegib-naive.
  * Cohort A2 - Participants had received prior vismodegib treatment.
* Cohort B - 200 mg itraconazole (as 100 mg twice daily, for up to 4 months). The objective of this cohort is to assess the anti-cancer efficacy of lower-dose extended treatment.
* Control Group - Tumors from untreated participants.

ELIGIBILITY:
INCLUSION CRITERIA

* At least one BCC tumor (greater than 4 mm in diameter) at any skin location, to be biopsied and surgically removed.
* Had at least one liver function test [eg, aspartate aminotransferase (AST), alanine aminotransferase (ALT)] with normal results in the last year.
* Consent to research use of their BCC tissue.
* Cohort A or B: Willing to take itraconazole during the 2 to 3 weeks between biopsy and surgical removal of BCC

EXCLUSION CRITERIA

* History or current hepatitis or other liver disease.
* Currently taking systemic medications that would affect BCC tumors (oral retinoids) or metabolism of itraconazole (anti-convulsants, corticosteroids)
* History or current evidence of malabsorption or liver disease within the one year prior to enrollment.
* History or current evidence of hyperthyroidism increasing metabolism of itraconazole
* Unable to attend to 2nd study visit at Stanford for Mohs surgical excision
* Current immunosuppression disease (cancer, autoimmune disease)
* Receiving immunosuppressive drugs
* Pregnant
* Lactating
* Any female actively trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Y Tang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim DJ, Kim J, Spaunhurst K, Montoya J, Khodosh R, Chandra K, Fu T, Gilliam A, Molgo M, Beachy PA, Tang JY. Open-label, exploratory phase II trial of oral itraconazole for the treatment of basal cell carcinoma. J Clin Oncol. 2014 Mar 10;32(8):745-51. doi: 10.1200/JCO.2013.49.9525. Epub 2014 Feb 3. PMID 24493717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Cohort A enrolled at the Stanford University Medical Center (SUMC). Subjects participated in biopsy studies.
  * Cohort B was enrolled and participated at the Universidad Catolica de Chile. No biopsy studies were conducted for these participants.
  * Untreated Control cohort was enrolled at SUMC. Subjects participated in biopsy studies.
Groups:
- Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve): Oral itraconazole 400 mg as 200 mg twice daily, for 1 month, for participants without prior vismodegib treatment (vismodegib-naïve) and more than 1 lesion at baseline.
- Cohort A2 - Itraconazole 400 mg (Prior Vismodegib): Oral itraconazole 400 mg as 200 mg twice daily, for 1 month, for participants with prior vismodegib treatment, and more than 1 lesion at baseline.
- Untreated Control: Participants otherwise eligible but unwilling to take itraconazole were enrolled onto the control arm of the study and received no treatment
Period: Overall Study
Arm/Group | Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg | Untreated Control
Started | 12 | 3 | 4 | 10
Completed | 9 | 3 | 4 | 10
Not Completed | 3 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with one or more BCC tumors measuring 4 mm or greater in diameter were enrolled.
Units Other Than Participants: Basal cell carcinoma lesions
Groups:
- Cohort B - Itraconazole 200 mg (Vismodegib-naïve): Oral itraconazole 200 mg as 100 mg twice daily, for up to 3 months treatment. All Cohort B participants were vismodegib-naïve.
- Total: Total of all reporting groups
Arm/Group | Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) | Untreated Control | Total
Number analyzed (Participants) | 12 | 3 | 4 | 10 | 29
Number analyzed (Basal cell carcinoma lesions) | 68 | 8 | 14 | 11 | 101
Age, Continuous [Mean (Full Range); unit: years] | 62.2 [44 to 85] | 57.7 [55 to 62] | 61.7 [51 to 78] | 68.5 [53 to 81] | 65.35 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 2 | 6
  Male | 9 | 3 | 3 | 8 | 23
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 0 | 10 | 25
  Chile | 0 | 0 | 4 | 0 | 4
Number of Tumor Lesions at Baseline [Count of Participants; unit: Participants]
  1 Tumor Lesion at Baseline | 8 | 3 | 0 | 10 | 21
  > 1 Tumor Lesion at Baseline | 4 | 0 | 4 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ki67 Tumor Proliferation Biomarker
Description: Percent change in Ki67 tumor proliferation biomarker was assessed at baseline and after 1 month of treatment, for Cohort A1 (vismodegib-naïve participants receiving 400 mg as 200 mg twice daily) vs control patients. The outcome is expressed as the % change from baseline of cells with a positive signal after staining for Ki67.
  * Paired analysis of tumors shows percent change between baseline (prior to treatment) and post itraconazole treatment in individual patients, & is reported as the mean of the changes observed for those lesions for which both baseline and treated valued are available.
  * Unpaired analysis shows percent change between individual tumors from control patients and itraconazole treated patients, and is reported as the change in mean of the group of baseline basal cell carcinoma (BCC) lesion measurements and the group of treated BCC lesion measurements.
Time Frame: 1 month
Population: Ki67 tumor proliferation biomarker assessment was not performed for Cohorts A2 (itraconazole 400 mg & prior vismodegib) and B (itraconazole 100 mg twice daily).
Measure: Mean (Standard Deviation); unit: Mean percent change
Units Other Than Participants: Basal Cell Carcinoma (BCC) lesions
Arm/Group | Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) | Untreated Control
Number analyzed (Participants) | 8 | 0 | 0 | 10
Number analyzed (Basal Cell Carcinoma (BCC) lesions) | 31 | 0 | 0 | 23
Mean percent change
  Unpaired Analysis: number analyzed (Basal Cell Carcinoma (BCC) lesions) | 20 | 0 | 0 | 23
  Unpaired Analysis | 18 (17) |  |  | 0 (15)
  Paired Analysis: number analyzed (Basal Cell Carcinoma (BCC) lesions) | 16 | 0 | 0 | 23
  Paired Analysis | -19 (15) |  |  | 13 (12)
Statistical Analysis 1: Comparison: Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve); Percent change in Ki67 tumor proliferation biomarker from baseline to 1 month, for Cohort A1 (vismodegib-naive patients, n = 8). Paired analysis of tumors shows percent change between baseline (prior to treatment) and post-itraconazole treatment in individual patients. % change was calculated from the difference between the mean of baseline Ki67 levels and the mean Ki67 levels after 1 month of treatment; Test type: Other; p = 0.04, t-test, 2 sided
Statistical Analysis 2: Comparison: Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve); Percent change in Ki67 tumor proliferation biomarker - baseline vs 1 month - Cohort A, vismodegib-naive (n = 8) vs control patients Unpaired analysis shows percent change between individual tumors from control patients and itraconazole treated patients. % change was calculated from the difference between the mean of baseline Ki67 levels and the mean Ki67 levels after 1 month of treatment; Test type: Other; p = 0.079, t-test, 1 sided
Statistical Analysis 3: Comparison: Untreated Control; Percent change in Ki67 tumor proliferation biomarker - baseline vs 1 month - control patients Paired analysis of tumors shows percent change between baseline and after 1 month in individual patients. % change was calculated from the difference between the mean of baseline Ki67 levels and the mean Ki67 levels after 1 month; Test type: Other; p = 0.652, t-test, 2 sided

2. Secondary Outcome: Change of GLI1 Tumor Biomarker
Description: Tumor biomarker GLI1 (glioma-associated oncogene 1), part of the Hedgehog (HH) pathway, was assessed in vismodegib-naïve participants at baseline and after 1 month of treatment by quantitative polymerase chain reaction (qPCR). The relative expression of the biomarker was measured as the fold increase of GLI1 expression compared to that of housekeeping gene hypoxanthine-guanine phosphoribosyltransferase (HPRT), and the outcome was assessed as the percent change from the mean of the pre-treatment measurements to the mean of the post-treatment measurements. A negative mean indicates an overall reduction in GLI1 expression.
Time Frame: 1 month
Population: Analysis conducted for Cohorts A1 - Itraconazole 400 mg (Vismodegib-naive) and A2 - Itraconazole 400 mg (Prior Vismodegib) only. GLI1 tumor biomarker assessment was not performed for the Cohort B (100 mg twice daily); or Control Group.
Measure: Mean (Standard Deviation); unit: Percent change
Units Other Than Participants: Basal Cell Carcinoma (BCC) lesions
Groups:
- Cohort B - Itraconazole 200 mg (Vismodegib-naïve): Oral itraconazole 200 mg as 100 mg twice daily, for up to 3 months treatment. All Cohort B participants were vismodegib-naïve, and had more than 1 lesion at baseline.
- Untreated Control: Participants otherwise eligible but unwilling to take itraconazole were enrolled onto this study control arm, and received no treatment.
Arm/Group | Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) | Untreated Control
Number analyzed (Participants) | 3 | 3 | 0 | 0
Number analyzed (Basal Cell Carcinoma (BCC) lesions) | 18 | 6 | 0 | 0
Percent change | -40.3 (35.6) | -16.2 (13.1) |  |
Statistical Analysis 1: Comparison: Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve); Percentage change in GLI1 messenger RNA (mRNA) expression Paired analysis of tumors shows percent change between baseline (prior to treatment) and post itraconazole treatment in individual patients. % change was calculated from the difference between the mean of baseline Gli levels and the mean Gli level after 1 month of treatment; Test type: Other; p = 0.028, t-test, 2 sided; Wilcoxon signed rank test

3. Secondary Outcome: Tumor Size
Description: Tumor size was assessed by caliper measurement of the longest perpendicular diameters before and after itraconazole treatment, and determination of tumor area by multiplication of the measurements for each tumor. The outcome is expressed as the mean percent change in tumor area from baseline, with standard deviation. A negative value indicates a reduction in size.
Time Frame: Up to 3 months
Population: Change in tumor area was assessed for only for Cohort A1 or B participants who had > 1 basal cell carcinoma (BCC) tumor (42 and 14 lesions respectively). No Cohort A2 participants had > 1 BCC tumor. No data were collected from untreated patients.
Measure: Mean (Standard Deviation); unit: Mean percent change
Units Other Than Participants: Basal Cell Carcinoma (BCC) lesions
Arm/Group | Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) | Untreated Control
Number analyzed (Participants) | 4 | 0 | 4 | 0
Number analyzed (Basal Cell Carcinoma (BCC) lesions) | 42 | 0 | 14 | 0
Mean percent change | -25.4 (21.8) |  | -20 (24.4) |
Statistical Analysis 1: Comparison: Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) vs Cohort B - Itraconazole 200 mg (Vismodegib-naïve); Only tumors from 4 patients from cohort A (n = 42 BCCs) and all tumors from the 4 patients (n = 14 BCCs) in cohort B were observed for tumor size change. Percent change in tumor area from both cohorts (eight patients total with 57 tumors) was calculated only; Test type: Other; Mean Difference (Final Values) = 24, 95% CI 2-sided [18.2 to 30]
Statistical Analysis 2: Comparison: Cohort A1 - Itraconazole 400 mg (Vismodegib-naïve) vs Cohort B - Itraconazole 200 mg (Vismodegib-naïve); Average tumor size reductions were compared between Cohort A1 and Cohort B; Test type: Other; p = 0.435, t-test, 1 sided

4. Secondary Outcome: Tumor Response
Description: The following criteria for basal cell carcinoma (BCC) tumor response were used.
  * Complete response (CR) means no visible evidence of any lesion consistent with BCC
  * Partial response (PR) means less than CR, but there was a visible decrease in BCC tumor size
  * No response (NR) / Stable Disease (SD) means no visible decrease in BCC tumor size
  * Progressive disease (PD) means an increase in size or number of BCC tumor lesions
  Treatment assessment was conducted on the basis of lesion photographs by a dermatologist investigator who was blinded to the assigned treatment.
Time Frame: End of treatment period: 1 month (Cohort A) or 2.3 months (mean for Cohort B)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A1 - Itraconazole 400 mg, (Vismodegib-naïve): Oral itraconazole 400 mg as 200 mg twice daily, for 1 month, for participants without prior vismodegib treatment (vismodegib-naïve) and more than 1 lesion at baseline.
Arm/Group | Cohort A1 - Itraconazole 400 mg, (Vismodegib-naïve) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) | Untreated Control
Number analyzed (Participants) | 4 | 3 | 4 | 10
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Partial Response (PR) | 4 | 0 | 0 | 0
  No Response (NR) / Stable Disease (SD) | 0 | 3 | 4 | 10
  Disease Progression (PD) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2.3 months (average)
Description: All patients treated with itraconazole were monitored for adverse events ≥ Grade 2. Only adverse events (AEs) grade 2 or greater were collected and reported.
Groups:
- Cohort A1 - Itraconazole 400 mg +/- Prior Vismodegib; Cohort A2 - Itraconazole 400 mg (Prior Vismodegib): Oral itraconazole 400 mg as 200 mg twice daily, for 1 month.
Arm/Group | Cohort A1 - Itraconazole 400 mg +/- Prior Vismodegib | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/12 | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 - Itraconazole 400 mg +/- Prior Vismodegib (N=12) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) (N=3) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) (N=4)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — One grade 4 congestive heart failure occurred in a patient who had undiagnosed heart disease from prior adriamycin treatment for Hodgkin lymphoma 20 years previously.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 - Itraconazole 400 mg +/- Prior Vismodegib (N=12) | Cohort A2 - Itraconazole 400 mg (Prior Vismodegib) (N=3) | Cohort B - Itraconazole 200 mg (Vismodegib-naïve) (N=4)
Grade 2 Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No